CLINICAL TRIAL: NCT03672370
Title: Alloclassic® Variall® Cup Ceramic Bearing System in Total Hip Arthroplasty A Multi-center, Prospective, Non-controlled Post Market Surveillance Study
Brief Title: PMCF Study on the Safety and Performance of the Alloclassic Variall Cup Ceramic Bearing System in Total Hip Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: Study terminated as CE marks of the devices used have not been renewed.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2014-03H.1
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-11

CONDITIONS: Avascular Necrosis; Osteoarthritis; Inflammatory Arthritis; Posttraumatic Arthritis
Keywords: Total hip arthroplasty; Medical device; Performance; Safety; Hip prosthesis
MeSH Terms: conditions — Osteonecrosis; Osteoarthritis; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alloclassic® Variall® Cup: Subjects who received the Alloclassic® Variall® Cup Ceramic Bearing System

SUMMARY:
The study is a multicenter, prospective, non-randomized, non-controlled consecutive cohort post-market clinical follow-up study.

DETAILED DESCRIPTION:
The objectives of this study are to obtain survival and outcomes data on the Alloclassic® Variall® Cup in combination with the BIOLOX® delta Taper Liner and a BIOLOX® delta Femoral Head used in primary total hip arthroplasty. This will be done by analysis of standard scoring systems, radiographs and adverse event records.

Two sites are involved in this study, enrolling a total of 100 patients for the study. All subjects were required to participate in the Informed Consent Process.

ELIGIBILITY:
Inclusion Criteria:

* Patient is skeletally mature.
* Patient qualifies for primary unilateral or bilateral total hip arthroplasty (THA) based on physical exam and medical history including the following:

  * Avascular necrosis (AVN)
  * Osteoarthritis (OA)
  * Inflammatory arthritis
  * Post-traumatic arthritis
* Patient has no history of previous prosthetic replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.) of the affected hip joint(s).
* Patient has a Harris Hip Score <70 in the affected hip
* Patient is willing and able to provide written informed consent.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the Ethics Committee approved informed consent.

Exclusion Criteria:

* The patient is:

  * A prisoner
  * Mentally incompetent or unable to understand what participation in the study entails
  * A known alcohol or drug abuser
  * Anticipated to be non-compliant.
* The patient has a neuromuscular disorder, vascular disorder or other conditions that could contribute to prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* The patient has a neurologic condition in the ipsilateral or contralateral limb which affects lower limb function.
* The patient has a known history of systemic disease that could affect his/her safety or the study outcome.
* The patient is known to be pregnant.
* The patient is unwilling or unable to give informed consent, or to comply with the follow-up program.
* The patient is not having any other investigational drug or device simultaneously.
* The patient has an active or latent infection in or about the affected hip joint or an infection distant from the hip joint that may spread to the hip hematogenously.
* The patient has insufficient bone stock to fix the component. Insufficient bone stock exists in the presence of metabolic bone disease (i.e. clinical relevant osteoporosis), cancer, and radiation. Note: Dual Energy X-ray Absorptiometry (DEXA) may be used to assess the presence of adequate bone stock.
* The patient has osteoradionecrosis in the operative hip joint
* The patient has a known sensitivity or allergic reaction to one or more of the implanted materials.
* The patient has known local bone tumors in the operative hip.
* The patient is Grade III obese with a Body Mass Inldex (BMI) > 40.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of a primary Total Hip Arthroplasty which receive the Alloclassic® Variall® Cup in combination with a BIOLOX ® delta Taper Liner and a BIOLOX ® delta Femoral Head
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (2):
- Austria (2):
  - Herz-Jesu Krankenhaus, Vienna
  - Orthopädisches Spital Speising GmbH, Vienna

RESULTS

PARTICIPANT FLOW:
Groups:
- Alloclassic Variall Cup: Subjects who received the Alloclassic Variall Cup Ceramic Bearing System
Period: Overall Study
Arm/Group | Alloclassic Variall Cup
Started | 89 (11 hips did not receive the study devices acc. to the protocol and therefore had to be excluded.)
Completed | 42
Not Completed | 47

BASELINE CHARACTERISTICS:
Arm/Group | Alloclassic Variall Cup
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 89
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success Will be Based on the Harris Hip Scoring System
Description: The Harris Hip Score (HHS) was developed for the assessment of the results of hip surgery, and is intended to evaluate various hip disabilities and methods of treatment in an adult population. The domains covered are pain, function, absence of deformity, and range of motion. The score has a minimum of 0 points and a maximum of 100 points.
  Clinical success will be defined as a modified Harris Hip score of > 80 that included a rating of 'mild', or 'no pain'; a failure will be defined as a modified Harris Hip score < 80.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alloclassic Variall Cup
Number analyzed (Participants) | 42
score on a scale | 92.6 (8.9)

2. Primary Outcome: Percentage of Participants Who Survived According to the Survival Analysis With the Kaplan Meier (K-M) Estimate
Description: Endpoint revision of any investigational device for any reason attributable to any investigational device
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alloclassic Variall Cup
Number analyzed (Participants) | 89
percentage of participants | 98.63 [90.67 to 99.81]

3. Secondary Outcome: Oxford Hip Score
Description: The purpose of the Oxford Hip Score (OHS) is to assess the outcome after total hip arthroplasty by measuring cases' perceptions in adjunction to surgery. The OHS assesses pain (6 items) and function (6 items) of the hip in relation to daily activities such as walking, dressing, sleeping, etc.
  The scoring is the following: 0-4 (worst to best) with overall scores ranging from 0-48 where 48 represents the best score
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alloclassic Variall Cup
Number analyzed (Participants) | 42
score on a scale | 44.7 (7.9)

4. Secondary Outcome: EQ-5D
Description: The EQ-5D questionnaire comprises two parts. For the first part, respondents are asked to tick boxes to indicate the level of problem on each of the five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). In total, there are three levels per dimension (no problems/no pain/not worried, some problems/some pain/a bit worried, a lot of problems/a lot of pain/very worried). Responses are coded as single-digit numbers expressing the severity level selected in each dimension. The digits for the five dimensions are combined in a 5-digit code.
  The second part of the questionnaire is the EQ Visual Analogue Scale. This captures the respondent's overall assessment of their health from 0 (worst health imaginable) to 100 (best health imaginable).
  The results from both parts are indexed, weightened and pulled together. The final score lies between 1 for full health and 0 for death. Values less than 0 are possible considered to be worse than death.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alloclassic Variall Cup
Number analyzed (Participants) | 42
score on a scale | 0.9 (0.2)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Alloclassic Variall Cup
All-Cause Mortality (participants affected / at risk) | 1/89
Serious Adverse Events (participants affected / at risk) | 7/89
Other Adverse Events (participants affected / at risk) | 2/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alloclassic Variall Cup (N=89)
Infection, revision required (Infections and infestations) | 2
Periprosthetic fractures, revision required (Musculoskeletal and connective tissue disorders) | 2
Lung cancer, unknown treatment (Respiratory, thoracic and mediastinal disorders) | 1
Traumatic event at outpatient rehab, surgical fragment fixation (Musculoskeletal and connective tissue disorders) | 1
Death, unknown reason, no relation to device (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alloclassic Variall Cup (N=89)
femoral implant loosening (Musculoskeletal and connective tissue disorders) | 1 — A patient mentioned a femoral implant loosening at the phone, which was treated in another hospital, however was not able to provide any further details. The patient asked for discontinuation of the study.
Pain in hip when sitting down, radiating to the knee (Musculoskeletal and connective tissue disorders) | 1 — Patient reported slight pain when sitting down, radiating to the knee. The pain is tolerated and no further treatment is required at the moment. No further information to this case were available.

LIMITATIONS AND CAVEATS:
Early termination of the study, many withdrawals of patients as they felt good and did not see the necessarity to come back to the follow-up visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT03672370/Prot_SAP_000.pdf